CLINICAL TRIAL: NCT06069089
Title: Assiut University, Pediatrician Department
Brief Title: Bone Denisty Change in Children With Beta Thalassemia Major
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marwa Hassan Abdelhamed Hassan (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Marwa Hassan Abdelhamed Hassan, Assiut university , pediatrician department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Thalassemia major in children
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Evaluate Bone Denisty Changes in Children With Beta Thalassemia Major
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled beta thalassemia major: Controlled beta thalassemia major Hb>9g/dl , serum ferritin <500ng/ml
  Interventions: Radiation: Dexa scan
- Uncontrolled beta thalassemia major: Uncontrolled beta thalassemia major Hb<9g/dl , serum ferritin >500ng/ml
  Interventions: Radiation: Dexa scan

INTERVENTIONS:
Radiation: Dexa scan — No intervention

SUMMARY:
Bone denisty changes in children with beta thalassemia major

DETAILED DESCRIPTION:
Beta Thalassemia major (TM) is a hereditary disease caused by defective Beta globin chain synthesis, resulting in abnormal as well as a decreased quantity of globin chains, ineffective erythropoiesis, haemolysis and increased red blood cell turnover (Cooley, etal, 1927). described the first patient with anemia, splenomegaly, cranial & facial bone enlargement. Pathophysiology of bone denisity changes in beta thalassemia major Several studies had been previously evaluated; shown that multiple factors may act in concert to produce bone disease in beta thalassemia major (TM) including bone marrow expansion (Shamshirsaz, etal, 2003). hypogonadism (Anapliotou,Saka&Jensen,1998), defective growth hormone-insulin-like growth factor-1 (GH-IGF-1) axis (Soliman,etal,1998), altered pattern of cytokines (Morabito,etal,2007), iron deposit in bone ((Bordat,etal,1993),deferoxamine bone toxicity (Chan ,etal, 2002),and vitamin D deficiency (Dandona, etal, 1987). Some of these pathogenic factors, directly and/or indirectly, affect osteoblastic population, leading to depressed bone formation, while others often increase osteoclastic bone resorption.

Complications of transfusion dependent poorly controlled beta thalassemia major are;(1)-Osteoprosis; Iron overload impairs osteoid maturation and inhibits local mineralization to form focal osteomalacia. In addition, integration of iron in calcium hydroxyapatite affects the growth of crystals, which causes mineralization failure (Chan, etal, 2002), defective growth hormone-insulin-like growth factor-1 (GH-IGF-1) axis (Soliman, etal, 1998),altered pattern of cytokines (Morabito,etal, 2007), iron deposit in bone (Bordat, etal, 1993), deferoxamine bone toxicity (Chan, etal,2002). and vitamin D deficiency (Dandona, etal, 1987). (2)-Fractures; The introduction of red blood cell transfusion and concomitant iron chelation therapy has led to improved bone health through various mechanisms. It leads to a reduction in medullary expansion and cortical bone thinning, the reduced incidence of hypogonadism, and a reduction in other endocrine complications such as hypoparathyroidism and metabolic disorders that predispose to low bone density and fractures( Multicentre study, italian working group 1995). Z-score of bone density will be calculated. Z score is the preferred parameter in children. which is calculated as the number of standard deviations above or below the mean for the patient's age, sex,

ELIGIBILITY:
Inclusion Criteria:

- Patient diagnosed as B thalassemia major of both sexes, age range from 10-18 year, who are poorly controlled on frequant blood transfusion. The patient who doesn't have Hb level from 9-10 g/dl, in almost always less than 9 g/dl.

Exclusion Criteria:

* Known metabolic bone disease. Less than 10 year or more than 18 year. Bone disease Other than hemolytic anemia.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with beta thalassemia major with transfusion dependent
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate bone denisty in children with beta thalassemia major | One year
  To evaluate bone denisty in transfusion dependent beta thalassemia major & its relation to serum minerals &vit D To evaluate bone denisity in transfusion dependent beta thalassemia major & its relation to serum minerals &vit D To evaluate bone denisity in transfusion dependent beta thalassemia major &its relation to serrum minerals &vitD

REFERENCES:
- [Background] Gaudio A, Morabito N, Catalano A, Rapisarda R, Xourafa A, Lasco A. Pathogenesis of Thalassemia Major-associated Osteoporosis: A Review with Insights from Clinical Experience. J Clin Res Pediatr Endocrinol. 2019 May 28;11(2):110-117. doi: 10.4274/jcrpe.galenos.2018.2018.0074. Epub 2018 Jul 11. PMID 29991466